CLINICAL TRIAL: NCT06371469
Title: The Effect of the Against to Cancer Health Behavior Program Applied to Mothers of Intellectual Disabled Children on Cancer Screenings and Preventive Health Behaviors: Nonrandomized Controlled Study
Brief Title: Program of Health Behaviour Against to Cancer (PHeBAC)
Acronym: PHeBAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Habibe ÖZÇELİK, Lecturer Dr, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KAEK-769
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cancer Prevention; Health Behavior; Disability, Intellectual; Parents; Cancer Screening; Experimental Study Designs; Mothers; Disabilities Mental
MeSH Terms: conditions — Health Behavior; Intellectual Disability | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Mothers participating in the research will not know that they are in the intervention or control group. The data of the research will be collected by an independent investigator. In addition telephone support during the research process will be provided by the independent investigator, too
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PHeBAC is an acronym that defines multi-interventions to health behaviour against cancer.
  The intervention group will receive PHeBAC with multiple interventions including education, guidance, counseling, and case management in line with the 12 European Codes Against Cancer to reduce cancer risk. The PHeBAC interventions will be 8 weeks long, with two face-to-face and three telephone interviews.
  The first and the 4th week will be face-to-face with two different sessions of 45 minutes each; the 2nd, 6th, and 8th weeks will be phone calls of 15 minutes each.
  Interventions: Behavioral: PHeBAC
- Control Group (Active Comparator): The active control group will be given brochures from the Ministry of Health on cancer prevention and cancer screening recommendations and their questions will be answered.
  Contact information of the researchers will be given and they will be told that they can call if they have any questions.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: PHeBAC — Multi-interventions to health behaviour against cancer in mothers of Intellectual Disabled Children
  Other Names: Intervention Group
  Arms: Experimental
Behavioral: Control Group — Providing brochures from the Ministry of Health, answering questions and providing the researcher's phone number
  Arms: Control Group

SUMMARY:
The European Code Against Cancer contains 12 recommendations to reduce the risk of cancer. It is estimated that about half of all cancers could be prevented if all recommendations are followed.

The aim of this study was to evaluate the effectiveness of the Program of Health Behaviour Against Cancer (PHeBAC) applied to mothers of children with intellectual disabilities in increasing the participation of mothers and their children with intellectual disabilities in cancer screenings and their health behaviors against cancer. The goal is to improve the preventive health behaviors of children with intellectual disabilities and their mothers against cancer and to increase the rate of participation in cancer screenings. Specific targets are; not smoking and not being exposed to smoking, increasing physical activity, healthy nutrition, limiting alcohol consumption, protection from sunlight, HPV vaccination and increasing participation in breast, cervical and colorectal cancer screenings.

DETAILED DESCRIPTION:
Intervention Group: Program of Health Behaviour Against Cancer (PHeBAC): PHeBAC is an 8-week program consisting of five interviews, two face-to-face and three by telephone.

Face-to-face training will be provided in two different sessions of 45 minutes each in the first and 4th weeks, and telephone interviews of 15 minutes each in the 2nd, 6th and 8th weeks.

Each planned intervention will be organized by taking the opinions of experts working in this field. In addition, expert opinions will be taken for the content of the presentation of face-to-face individual trainings to the intervention group.

The pre-tests of the study will be collected just before the training in week 0 and the post-tests will be collected in week 9. Data collection forms will be filled in by the participants under the supervision of the researcher.

Intervention to be applied to the Control Group: Participants in the active control group will be invited for a face-to-face interview and the pretests will be completed by the participants under the supervision of the researcher. After the pre-tests are taken, the participants will be informed about the brochure of the Ministry of Health, which includes cancer prevention recommendations and cancer screening recommendations, and the content of the brochure. The contact information of the researchers will be given and they will be told that they can call if they have any questions. The post-tests will be completed in the ninth week. Data collection forms will be completed by the participants under the supervision of the researcher.

The data of the study will be evaluated using "the Health Behaviors and Participation in Cancer Screenings Data Collection Form developed by the researchers", "Healthy Lifestyle Behaviors Scale II-Physical Activity and Nutrition Sub-Factors", "Sun Protection Behavior Scale". IBM SPSS 23 and Gpower programs will be used for statistical analysis of the data obtained from the study. The distribution of the data will be evaluated with Skewness and Kurtosis. For continuous data showing normal distribution, t test in two dependent groups, Student t test in two independent groups, One-way ANOVA test will be performed. For categorical data, McNemar test in two dependent groups and chi-square test in two independent groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Those who have at least one intellectual disabled child receiving education at Special Education Application Center schools,

Exclusion Criteria:

* Caregivers other than the mother of the intellectual disabled child
* Mothers who are being followed up with a diagnosis of breast, cervix or colorectal cancer

Disqualification Criteria:

* Mothers in the PheBAC group who do not continue with the telephone meetings after the face-to-face interview

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers of intellectual disabled children will be included.
Enrollment: 46 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Health Behaviors and Participation in Cancer Screenings Data Collection Form | 8 weeks
  Developed by the researchers in line with the recommendations of the European Code Against Cancer. It includes information on smoking, secondhand smoke, alcohol use, HPV vaccination and cancer screenings.
Healthy Life Style Behaviors Scale II (Physical Activity and Nutrition Sub-Factors) | 8 weeks
  The scale consists of six sub-factors and two sub-factors, physical activity and nutrition, will be used. All items of the scale are positive. As the score increases, the level of physical activity and nutrition increases. The physical activity sub-factor consists of 8 items and the nutrition sub-factor consists of 9 items. The 4-point Likert scale is accepted as never (1), sometimes (2), frequently (3), and regularly (4).
Sun Protection Behavior Scale | 8 weeks
  It examines the sun protection behavior of the individual when the sun exposure time is more than 15 minutes. The scale consists of three sub-factors: regular sun avoidance, sunscreen use and hat use. All items of the scale are positive. As the score increases, sun protection behaviors increase. Sun avoidance consists of three items, sunscreen use consists of three items and hat use consists of two items. On a 5-point Likert scale, (1) is considered as never, (2) rarely, (3) sometimes, (4) usually and (5) always.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe OZCELIK, PhD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No